CLINICAL TRIAL: NCT05113823
Title: In Situ Simulation Training for a Better Interprofessional Team Performance in Transferring Critically Ill COVID-19 Patients: A Prospective Randomized Control Trial
Brief Title: In Situ Simulation Training in Transferring Critically Ill COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IndonesiaUAnes122
Record Dates: First submitted 2021-10-25; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Simulation of Physical Illness; COVID-19 Respiratory Infection
Keywords: In Situ Simulation; Intreprofessional Training; High Fidelity Mannequin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fidelity Simulator (Active Comparator): Subjects will receive training using high fidelity simulator
  Interventions: Procedure: Simulation Training
- Low Fidelity Simulator (Active Comparator): Subjects will receive training using low fidelity simulator
  Interventions: Procedure: Simulation Training

INTERVENTIONS:
Procedure: Simulation Training — Simulation Training using High and Low Fidelity Simulator

SUMMARY:
This study aimed to determine the role of in situ simulation training during a pandemic by using standard and high-fidelity mannequins to improve interprofessional communication, skills, and teamwork in transferring critically ill COVID-19 patients.

DETAILED DESCRIPTION:
Fourty subjects were randomly allocated into two large groups, the High Fidelity Simulator group and the Low Fidelity Simulator group. Each group was divided into small groups, consist of 2 doctors and 3 nurses. All subjects underwent the same interactive lectures, and two sessions of in-situ simulation according to their assign group. In-situ simulation and debriefing were performed by implementing appropriate personal protective equipment and social distancing. At the end of each simulation session, each group would underwent a debriefing session, which was performed by an experience instructor. The first simulation was aimed to teach participants skills and steps in transporting critically-ill COVID-19 patients according to the hospital check-list. While the second simulation was aimed to assess skills, team work and communication that participants had learned from the previous simulation, by using assessment tools that had been developed before. In addition to comparing each point in the assessment tool between the two groups, the points that had been earned were also added up to get the overall points for total skills, cooperation and communication score. At the end of the session, learner immediate feedback were also collected using an online feedback form, which provided accountability for attendance, content learning, and course evaluation feedback.

ELIGIBILITY:
Inclusion Criteria:

* in good physical condition
* had no history of involving in COVID-19 patients care
* willing to become study subject

Exclusion Criteria:

* doesn't want to become study subject

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
rate of interprofessional communication | within 3 months
  improvement of interprofessional communication in transferring critically ill COVID-19 patients
rate of skill | within 3 months
  improvement of skill in transferring critically ill COVID-19 patients
rate of team work | within 3 months
  improvement of team work in transferring critically ill COVID-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Derived] Manggala SK, Tantri AR, Sugiarto A, Sianipar IR, Prasetyono TOH. In situ simulation training for a better interprofessional team performance in transferring critically ill patients with COVID-19: a prospective randomised control trial. Postgrad Med J. 2022 Aug;98(1162):617-621. doi: 10.1136/postgradmedj-2021-141426. Epub 2022 Jan 31. PMID 35101969